CLINICAL TRIAL: NCT05496153
Title: The Clinical Effect of Adaptive Posture-balance Cardiac Rehabilitation Exercise on Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ting Li, Director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Balance-based rehabilitation
Record Dates: First submitted 2022-07-29; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Rehabilitation; Exercise Therapy; Balance Exercises; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiovascular diseases Patients (Experimental): Subjects were recruited from outpatients with CVDs, under 18 years of age. All pa-tients have been verified the willingness of participating before the experiment. Patients was excluded if having abnormal blood pressure response, unstable angina pectoris, acute heart failure, congenital heart disease, and severe musculoskeletal diseases limiting.
  Interventions: Behavioral: Adaptive posture-balance cardiac rehabilitation exercise

INTERVENTIONS:
Behavioral: Adaptive posture-balance cardiac rehabilitation exercise — The process of APBCRE consisted of four parts: breathing training and warm-up, aerobic exercise, resistance exercise, and flexibility exercise. The first part lasted for 5-15 minutes, based on balance exercise. The specific steps of balance exercise included stretching of upper limbs, legs, waist, and other parts. And the second part was generally moderate-intensity endurance exercise, thresholding for 60%-75% VO2max/kg metabolic equivalents (METs), 60%-70% maximum heart rate, rating of perceived exertion (RPE) Borg grade 12-13. The exercise duration of this part was usually 30 min. During the self-created APBCRE, the resistance exercise was carried out with the help of the body-building vehicle, and its power was adjusted based on danger assessment level and oxygen uptake at anaerobic threshold. The last part usually lasted for 5-10 min for each-level participants. The total exercise time for one session was generally 50-70 min.

SUMMARY:
The whole experiment included one-month APBCRE therapy and two assessments. The one-month APBCRE consisted of twelve exercise sessions, evenly three times per week. At baseline and after rehabilitation, participants underwent one assessment, including car-diopulmonary exercise testing (CPET), resting metabolic rate (RMR) detection, and quality of life questionnaire (QoL). The primary outcomes were exercise capacity measured by function parameters at anaerobic threshold (AT) and other CPET physiological indexes. The secondary endpoints were the RMR level and QoL score.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* With cardiovascular diseases

Exclusion Criteria:

* abnormal blood pressure response
* unstable angina pectoris
* acute heart failure
* congenital heart disease
* severe musculoskeletal diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
CPET | Baseline and immediately after the intervention, about one month
  Cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Quality of life | Baseline and immediately after the intervention, about one month
  Using 12-Item Short Form Survey questionnaire to assess the quality of life
RMR | Baseline and immediately after the intervention, about one month
  Resting metabolic rate

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Chest Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No